CLINICAL TRIAL: NCT00323986
Title: Azithromycin Treatment of Patients With Chronic Obstructive Pulmonary Disease (COPD) and Tracheostomy. Effects on Recurrent Respiratory Infections, Inflammatory Parameters and Bacterial Persistence
Brief Title: Azithromycin Treatment of Patients With Chronic Obstructive Pulmonary Disease (COPD) and Tracheostomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 39/2004
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2006-05-10 (Estimated); Status verified 2006-04

CONDITIONS: COPD; Tracheostomy
Keywords: COPD; tracheotomy; azithromycin; exacerbation; hospitalisation; exhaled breath condensate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Azithromycin; Pharmaceutical Preparations

INTERVENTIONS:
Drug: azithromycin (drug)

SUMMARY:
Aims of the study

* to evaluate the rate of enteric gram negative bacteria colonization in tracheotomised COPD patients
* to evaluate the effect of azithromycin long-term treatment on Pseudomonas aeruginosa colonization and colony counts, and on reduction of the number of exacerbations/hospitalisations, antibiotic courses and steroid use.
* to evaluate the Quality of Life of patients treated and not treated with azithromycin, using a validate Italian version of St George questionnaire
* to evaluate the rate of chronic colonization with atypical pathogens
* to evaluate the safety and tolerability of a long-term treatment with azithromycin, including a survey on possible bacterial antibiotic resistance pattern variations

DETAILED DESCRIPTION:
Methods. Study Design Prospective, randomised, multicentre study. Centers

* Dott. E. Guffanti, IRCCS INRCA Casatenovo, Varese Italy
* Prof. F. Blasi, Università degli Studi di Milano, IRCCS Ospedale Maggiore Milan Italy
* Dott, M. Confalonieri, Ospedale Trieste, Italy Patients

We plan to enrol 30 patients :

Inclusion criteria

* Age > 45 years
* Tracheotomy
* History of COPD demonstrated by pulmonary function tests
* Informed Consent Exclusion criteria

  * Allergy to macrolides
  * Life expectancy < 1 year

Exhaled breath condensate (EBC) The breath condensate samples is collected using a specially designed condensing chamber (Ecoscreen; Jaeger, Hoechberg, Germany). The exhaled air entered and left the chamber though one-way inlet and outlet valves, thus keeping the chamber closed. The subjects wear noseclips and breathed tidally through a mouthpiece connected to the condenser for ten minutes. Approximately 1 ml of the sampled material is transferred to 2-ml plastic tube and stored at -70°C.

Interleukin-6 assay Interleukin-6 concentrations in the breath condensate will be measured using a specific enzyme immunoassay kit (EIA) (Cayman Chemical, Ann Arbor, USA). The assay is directly validated by means of gas chromatography/mass spectrometry in order to obtain a high correlation (r=0.95) between known amounts of IL-6 and the concentration measured by the EIA. The detection limit of the assay was 1.5 pg/ml after a two-hour development period.

TNF alfa TNF-alfa serum levels will be measured by enzyme immunoassay (Cayman Chemical, Ann Arbor, USA)

Microbiology Quantitative culture of tracheal aspirate will be performed at steady state, every 3 months and at exacerbation. Molecular biology techniques for Streptococcus pneumoniae, Haemophilus influenzae, Moraxella catarrhalis, Pseudomonas aeruginosa, Chlamydia pneumoniae and Mycoplasma pneumoniae identification will be also applied on the same specimens.

Timetable Enrolment: between January 2004 and December 2005 Visits : Every 3 months and on each exacerbation/hospitalization a visit will be performed. Every month a phone call will be performed.

Follow-up: 12 months. End of the study : July 2006

Visit

1. Visit 1. A complete history will be recorded. Inclusion and exclusion criteria will be checked. Informed consent will be collected and QoL questionnaire completed. Tracheal aspirate will be performed and divided into two aliquots : one for the local microbiology lab for quantitative cultures, and one for central lab for bacterial detection by PCR (stored at -80°C). Exhaled breath samples will be obtained.
2. Follow-up visits. Every 3 months the patients will be recalled at the center and all Visit 1 procedures will be repeated. Number of exacerbations/hospitalisation will be recorded and QoL questionnaire completed.
3. Exacerbation/hospitalisation visit. In presence of symptoms deterioration patients will be instructed to contact the center for a visit. All Visit 1 procedures will be repeated.
4. End of the study visit. At the end of the 12 month follow-up all Visit 1 procedures will be repeated. Number of exacerbations/hospitalisation will be recorded and QoL questionnaire completed.

Treatment Patients will be randomised to receive usual care or usual care + Azithromycin 500 mg o.d. three day-a-week (Monday, Tuesday, Wednesday) for 6 months.

Outcome measures

* reduction of inflammatory cytokines in EBC
* reduction of colony counts/eradication of bacteria on bronchial aspirates
* reduction of number of exacerbations/hospitalisations
* reduction of steroids and antibiotics use
* Quality of life

ELIGIBILITY:
Inclusion Criteria:

* Age > 45 years Tracheotomy History of COPD demonstrated by pulmonary function tests Informed Consent

Exclusion Criteria:

* Allergy to macrolides Life expectancy < 1 year

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-10; Study Completion 2006-04

PRIMARY OUTCOMES:
reduction of number of exacerbations
reduction of number of hospitalisations

SECONDARY OUTCOMES:
reduction of colony counts/eradication of bacteria on bronchial aspirates
reduction of steroids and antibiotics use
reduction of inflammatory cytokines in EBC

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Blasi, MD, Principal Investigator — Istituto Malattie Respiratorie University of Milan Italy
Locations (3):
- Italy (3):
  - Istituto Nazionale di riposo e cura per anziani (INRCA), Casatenovo
  - Istituto Malattie Respiratorie University of Milan, Milan
  - University Hospital Trieste, Trieste

REFERENCES:
- [Derived] Blasi F, Bonardi D, Aliberti S, Tarsia P, Confalonieri M, Amir O, Carone M, Di Marco F, Centanni S, Guffanti E. Long-term azithromycin use in patients with chronic obstructive pulmonary disease and tracheostomy. Pulm Pharmacol Ther. 2010 Jun;23(3):200-7. doi: 10.1016/j.pupt.2009.12.002. Epub 2009 Dec 16. PMID 20025989